CLINICAL TRIAL: NCT00183352
Title: Reproductive Endocrine Function and Mood Over the Menstrual Cycle of Women Treated for Bipolar Disorder
Brief Title: Reproductive Function and Mood in Women With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Natalie Rasgon, Professor, Stanford University
Other Study IDs: R01MH066033 (NIH); R01MH066033 (NIH); SPO# 28571; DAHBR 96-BHC
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2009-04

CONDITIONS: Bipolar Disorder; Mental Health
Keywords: Women; Mood; Menarche; Menstruation
MeSH Terms: conditions — Bipolar Disorder; Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women with bipolar disorder
- 2: Women who are healthy controls

SUMMARY:
This study will determine the effect of medication for bipolar disorder on the reproductive function and whether mood changes occur during the menstrual cycle in women with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a serious condition that can have devastating effects on social and psychological functioning. Evidence suggests that medications for bipolar disorder may influence reproduction function among women. This study will determine reproductive function and mood changes in women who are currently on medication for bipolar disorder.

This study will comprise women with bipolar disorder and age- and body mass index (BMI)-matched healthy controls. Participants will have their reproductive function and mood changes assessed for 3 consecutive menstrual cycles. Daily, participants will report about their mood, sleep patterns, life events, and any psychiatric medications; this information will be entered into a computerized system named ChronoRecord. In addition, participants will measure their basal body temperature and collect their urine every morning to assess for ovulation. Blood collection will occur at study entry and between Days 3 and 6 of every menstrual cycle to determine levels of reproductive hormones. Participants will be asked to fast for 12 hours prior to every blood collection. During the first month of the study, an extra study visit will occur. Participants will undergo a physical exam for determination of excessive hair growth (hirsutism) and BMI. Additionally, insulin resistance will be measured, and participants will be asked to complete a questionnaire that will be used to determine their past and current menstrual function, as well as the reproductive and psychiatric history of their families.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Have been menstruating for at least 4 years prior to study entry
* Participants must be willing to travel to Stanford University at own expense for study visits

Inclusion Criteria for Bipolar Disorder Participants:

* Participants should have a diagnosis of Bipolar I, Bipolar II, or Bipolar not otherwise specified (NOS), and be under the treatment of a physician who can be contacted in case of an emergency
* Current treatment with any mood-stabilizing agent for a period of at least 3 months (e.g., divalproex sodium, lithium, other mood stabilizer, or atypical antipsychotic)

Inclusion Criteria for Healthy Controls:

* No past or present diagnosis of mental illness

Exclusion Criteria for All Participants:

* Current alcohol or substance abuse or dependence within 6 months prior to study entry
* Meets criteria for another DSM-IV Axis I disorder
* Contraceptive steroid use within 3 months prior to study entry
* Current use of medication that may affect steroid metabolism
* Menopausal
* Endocrine disease such as diabetes or hypothyroidism
* Uncontrolled medical illness
* History of long-term corticosteroid use
* Organic mood disorder
* Pregnancy or breastfeeding within 3 months prior to study entry

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women diagnosed with Bipolar Disorder, between 18-40 years of age, who are currently treated with a mood stabilizing agent for a period of at least 3 months and are not taking birth control pills currently. Participants must be willing to travel to Stanford University (near San Francisco, CA) at their own expense for study visits.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie L. Rasgon, MD, PhD, Principal Investigator — Department of Psychiatry and Behavioral Sciences, Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States